CLINICAL TRIAL: NCT00861120
Title: Panitumumab and Pegylated Liposomal Doxorubicin for Platinum-Resistant Epithelial Ovarian Cancer With Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Wild-type
Brief Title: Panitumumab and Pegylated Liposomal Doxorubicin for Platinum-Resistant Epithelial Ovarian Cancer With KRAS Wild-type
Acronym: PaLiDo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-007799-13
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Ovarian cancer; KRAS wildtype; Platinum resistant
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — liposomal doxorubicin; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — 40 mg/m2 on day 1 of a 28 days cycle
  Other Names: Caelyx
Drug: Panitumumab — 6 mg/kg on days 1 and 15 of a 28 days cycle
  Other Names: Vectibix

SUMMARY:
The purpose of this study is to investigate the response rate in platinum-resistant, KRAS wild-type, ovarian cancer patients who are treated with pegylated liposomal doxorubicin (Caelyx®) in combination with biological treatment panitumumab (Vectibix®).

DETAILED DESCRIPTION:
Patients with platinum-resistant recurrent ovarian cancer have few therapeutic options and the response rates are only 10-20% using non-cross-resistant chemotherapeutic agents.

New biologic agents in combination with chemotherapy or other treatment modalities may result in improvement in survival.

Recent results in colorectal cancer have clearly indicated that KRAS mutant tumors do not respond to treatment with EGFR inhibitors.

Panitumumab (ABX-EGF) is the first fully human monoclonal antibody specific to the EGF receptor. To date, panitumumab has been evaluated in combination with chemotherapy in patients with CRC, NSCLC, and SCCHN.

No previous studies have evaluated the effect of panitumumab in epithelial ovarian cancer based on KRAS mutation status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial primary ovarian, primary fallopian or primary peritoneal cancer. Stage I-IV.

  * A: First line treatment with a platinum containing regimen with either progression or no response during 1.line chemotherapy, or relapse within 6 months after end of 1. line chemotherapy, OR
  * B: Patients receiving second line with a platinum containing regimen with either progression or no response during second line chemotherapy, or relapse within 6 months after end of second line chemotherapy
* Maximum two prior lines of chemotherapy (both platinum-based)
* Age ≥ 18 years.
* Performance status 0-2.
* Measurable disease by CA125 GCIG criteria
* KRAS wild type
* Adequate bone marrow function, liver function, renal function and coagulation parameters (within 7 days prior to randomization):

  * WBC ≥ 3.0 x 109/l or neutrophils (ANC)≥ 1.5 x 109/l
  * Platelet count ≥ 100 x 109/l
  * Hemoglobin ≥ 9.7 g/dl (6 mmol/L)
  * Serum bilirubin ≤ 1.5 x UNL
  * Serum transaminases ≤ 2.5 x UNL in absence of liver metastases, or ≤ 5xUNL in presence of liver metastases
  * Serum creatinine ≤ 1.5 x UNL
  * Magnesium ≥ lower limit of normal
  * Calcium ≥ lower limit of normal
* Written informed consent

Exclusion Criteria:

* Prior treatment with chemotherapy or biological targeted treatment except 1. line chemotherapy with platinum or combination platinum/taxane (bevacizumab allowed as part of the 1. line treatment).
* Patients who have received (or are planning to receive) treatment with any other investigational agent, or who have participated in another clinical trial within 28 days prior to entering this trial.
* Pregnant or breast-feeding or planning to become pregnant within 6 months after end of treatment. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use acceptable and safe methods of contraception during and for 6 months following treatment
* Other present or previous malignancy except curatively treated cervical cancer, non-melanotic skin cancer or other cancer with minimal risk of relapse.
* CNS metastasis
* History of any chronic medical or psychiatric condition or laboratory abnormality that are not medically controlled or in the opinion of the Investigator may increase the risks associated with study drug administration. (e.g. diabetes, cardiac diseases, hypertension).
* Clinically significant cardiovascular disease ≤ 1 year before enrollment/randomization, including:

  * Myocardial infarction or unstable angina within 6 months of randomization.
  * New York Heart Association (NYHA) ≥ Grade 2 congestive heart failure. Even if medically controlled.
  * Poorly controlled cardiac arrhythmia despite Medication (patients with rate-controlled atrial fibrillation are eligible)
* Uncontrolled hypercalcemia (calcium level outside the upper limit of normal; antihypercalcemic treatment is allowed).
* Allergy to the ingredients of the study medication or to Staphylococcus Protein A
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months.

SECONDARY OUTCOMES:
Progression Free Survival | 6 months.
Overall survival | Up to 5 years
Toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, MD, DMSc, Study Chair — Vejle Hospital; Karina D. Steffensen, MD, PhD, Principal Investigator — Vejle Hospital
Locations (6):
- AGO Austria, Innsbruck, Austria
- Leuven University Hospital, Leuven, Belgium
- Denmark (3):
  - Aalborg Hospital, Aalborg
  - Herning Regional Hospital, Herning
  - Vejle Hospital, Dept. of Oncology, Vejle
- Lund University Hospital, Lund, Sweden